CLINICAL TRIAL: NCT06907966
Title: Digital Implementation Support Strategies for Caregiver Home Practice
Brief Title: Digital Support Strategies for Caregiver Home Practice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, JoannaKim@asu.edu, Assistant Professor, Arizona State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00014233; K01DA055118 (NIH)
Record Dates: First submitted 2025-02-18; First posted 2025-04-03 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acceptability; Feasibility Studies
Keywords: home practice; parenting; skills practice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Engaging Families App (Experimental): Participants in this arm will receive the Engaging Families home practice app
  Interventions: Behavioral: Engaging Families home practice app
- Active control app (Active Comparator)
  Interventions: Other: Scheduling app

INTERVENTIONS:
Behavioral: Engaging Families home practice app — The intervention is a smartphone application (or "app") that was developed to support caregiver home practice of intervention skills. The app was designed to support caregivers participating in the Bridges program, an evidence-based, family-based preventive intervention. Features of the app were developed to help caregivers overcome common barriers to practicing intervention skills at home.
  Arms: Engaging Families App
Other: Scheduling app — The Cozi Family Organizer is a smartphone application that will be given to caregivers randomized to the active control group. Cozi is a highly rated family organization app with features that include a family calendar, to do list, shopping list, and daily agenda. Cozi is available on Android and iPhone devices.
  Arms: Active control app

SUMMARY:
This project is a pilot trial of the Engaging Families home practice smartphone application (or "app") as an add on to a family-based prevention program. Although there are many evidence-based preventive interventions delivered to caregivers to prevent youth substance use and mental illness and promote youth positive family and youth outcomes, the impact of these interventions is often limited by low home practice of intervention skills among caregivers. The Engaging Families home practice app is a digital behavior change intervention that was developed to support caregivers in practicing intervention skills at home. Researchers will ask participants if the app was acceptable and feasible for daily use at home. Researchers may also compare how often caregivers who use the study app do home practice of intervention skills compared with caregivers who do not receive the home practice app but are encouraged to use an app to help schedule their activities.

DETAILED DESCRIPTION:
The goals of the current pilot trial are to examine the acceptability and feasibility of the Engaging Families home practice smartphone application (or "app"). The Engaging Families app was developed and designed to support families who are already enrolled in and participating in the family-based prevention program Bridges. Families will be assigned to either receive the Engaging Families home practice app or another app to support parents' home practice of skills that they learn during the Bridges program. Acceptability and feasibility as well as preliminary effects will be assessed via survey measures. Select participants will be invited to participate in a post-intervention interview to also assess acceptability and feasibility of the app intervention.

ELIGIBILITY:
Caregiver Inclusion Criteria:

* Informed consent
* Ownership and regular use of a smartphone
* English or Spanish language fluency
* Concurrent enrollment in the family-based EBI Bridges
* Parent of a child aged 11-17 years old

Caregiver Exclusion Criteria:

- Decline to download the home practice app on their personal smartphone.

Child Inclusion Criteria:

* Parent/guardian consent
* Informed assent
* Parent is enrolled in the study
* English reading ability at the 4th grade level or higher

Child Exclusion Criteria:

* No parent/guardian consent
* Parent/guardian is not enrolled in the study concurrently

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the intervention | Post-intervention, approximately 2-3 months post baseline
  Acceptability of the intervention will be assessed using the Acceptability of Intervention Measure (AIM). This measure was developed specifically to support assessing the acceptability of implementation of a new intervention. Psychometric properties of this measure were assessed in prior studies. The final measures exhibited discriminate content validity and acceptable model fit. See Weiner, B.J., Lewis, C.C., Stanick, C. et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Sci 12, 108 (2017). https://doi.org/10.1186/s13012-017-0635-3 for more information.
  The following items are rated on a 5-point Likert-type scale (Complete disagree to Completely agree):
  [This program] meets my approval. [This program] is appealing to me. I like [this program]. I welcome [this program].
Intervention Feasibility | Post-intervention, approximately 2-3 months post baseline
  Feasibility of the intervention will be assessed using the Feasibility of Intervention Measure (AIM). This measure was developed specifically to support assessing the feasibility of implementation of a new intervention. Psychometric properties of this measure were assessed in prior studies. The final measures exhibited discriminate content validity and acceptable model fit. See Weiner, B.J., Lewis, C.C., Stanick, C. et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Sci 12, 108 (2017). https://doi.org/10.1186/s13012-017-0635-3 for more information.
  The following items are rated on a 5-point Likert-type scale (Complete disagree to Completely agree):
  1. (THIS INTERVENTION) seems implementable.
  2. (THIS INTERVENTION) seems possible.
  3. (THIS INTERVENTION) seems doable.
  4. (THIS INTERVENTION) seems easy to use.
Home practice of skills | 3 times during the intervention, up to 8 weeks
  At Sessions 2, 3, and 4, parents will respond to three questions about their experience completing home practice on a 6-point Likert-type scale:
  How many times did you practice [the skill]? (0 = did no practice to 5+ times) How well are you able to use [the skill] with your teen? (0 = did not practice, 1 = not at all to 5 = very well) How helpful was it to use [the skill] with your teen? (0 = did not practice, 1 = not at all to 5 = very helpful)

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project details from NIH Reporter — https://reporter.nih.gov/search/lNMkL5SDUEaDlI9RxkqlRw/project-details/10886789